CLINICAL TRIAL: NCT01794715
Title: Is Routine Ultrasound Examination Performed by Nurses Useful in Heart Failure Patients at a Outpatient Clinic
Brief Title: Ultrasound by Nurses in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: LH-2013-1; Spl hjertesvikt (Other: Levanger Hospital)
Record Dates: First submitted 2013-02-13; First posted 2013-02-20 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure
Keywords: Heart failure; Nurse led; Outpatient clinic; Echocardiography; Pocket-size; Ultrasound
MeSH Terms: conditions — Heart Failure | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound performed by nurses (Experimental): Examinations including ultrasound examinations
  Interventions: Procedure: Ultrasound examination by nurses
- Ultrasound not performed (Active Comparator): Examinations not including ultrasound examinations, otherwise active
  Interventions: Procedure: Ultrasound examination by nurses

INTERVENTIONS:
Procedure: Ultrasound examination by nurses — Ultrasound examination performed by nurses. Focused examination of the pleural space and inferior vena cava.
  Other Names: Ultrasound

SUMMARY:
Cross-over study aimed to study the diagnostic and clinical impact of routinely adding a pocket-size ultrasound examination to traditional care at a outpatient heart failure clinic.

DETAILED DESCRIPTION:
Patient inclusion: Outpatient heart failure clinic. Patients are eligible for inclusion if the are referred with heart failure and concent to participate in the study. No other exclusion criteria other than no willing/able to give their concent.

Study population: Approximately 80 patients Intervention: All participants will undergo careful medical history, physical examination and blood tests led by nurses. All patients will be examined twice (by two nurses), one will routinely add ultrasound examination of the pleural space and the inferior vena cava to assess volume state, the other nurse will not perform ultrasound examination. Full cross-over design were nurses do ultrasound examinations at a random matter.

Patients will then be examined by echocardiography by experience cardiologist's echocardiographers. Outcome measures:Change in therapy after routinely performed ultrasound examinations vs controls, detection of volume state when performing ultrasound examinations compared to controls with cardiologist's echocardiographic examination as a gold standard.

Descriptive data of patients before, under and after examinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the outpatient heart failure clinic at the local hospital

Exclusion Criteria:

* Not able or not willing to concent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Treatment effect | 0 and 30 days and 6 months
  Change in treatment after routinely performed ultrasound vs no ultrasound performed.

SECONDARY OUTCOMES:
Quality of nurse performed ultrasound | 0 and 30 days and 6 months
  Validation of nurse driven ultrasound. Measures of detection of volume state and specific ultrasonographic measurements compared to reference method (cardiologist performer ultrasound).

OTHER OUTCOMES:
proBNP vs ultrasound | 0 and 30 days
  Study of which variable that best predicts the clinical treatment of the population

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Levanger Hospital, Nord-Trøndelag Health Trust, Levanger, Norway

REFERENCES:
- [Derived] Gundersen GH, Norekval TM, Graven T, Haug HH, Skjetne K, Kleinau JO, Gustad LT, Dalen H. Patient-reported outcomes and associations with pleural effusion in outpatients with heart failure: an observational cohort study. BMJ Open. 2017 Mar 20;7(3):e013734. doi: 10.1136/bmjopen-2016-013734. PMID 28320791
- [Derived] Gundersen GH, Norekval TM, Haug HH, Skjetne K, Kleinau JO, Graven T, Dalen H. Adding point of care ultrasound to assess volume status in heart failure patients in a nurse-led outpatient clinic. A randomised study. Heart. 2016 Jan;102(1):29-34. doi: 10.1136/heartjnl-2015-307798. Epub 2015 Oct 5. PMID 26438785